CLINICAL TRIAL: NCT04155333
Title: Effects of Non-Invasive Brain Stimulation on Soldiers' Cognitive and Functional Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Aeromedical Research Laboratory (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: USAARL 2018-002; M-10782
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Performance Enhancement
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized, sham-controlled, within-subjects design
Who Masked: Investigator
Masking Description: Subjects and the research team will both be blind to the stimulation condition delivered at each test session. Access will be limited to the study physicians, investigators, and device programmers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active anodal stimulation (Experimental): active anodal stimulation at F3, cathode placed on contralateral bicep
  Interventions: Device: Transcranial direct current stimulation
- Active cathodal stimulation (Experimental): active cathodal stimulation at F3, anode placed on contralateral bicep
  Interventions: Device: Transcranial direct current stimulation
- Sham stimulation (Sham Comparator): sham stimulation that will be counterbalanced between subjects such that half will receive sham stimulation configured as condition 1 (anode F3, cathode bicep) and half will receive condition 2 (cathode F3, anode bicep)
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct current stimulation (tDCS) is a form of non-invasive brain stimulation that stimulates the brain through the application of a low-intensity electrical current, typically ranging from 1 to 2 milliamps (mA), via electrodes placed on an individual's scalp. During the active stimulation sessions, 2 mA of stimulation will be applied for 30 minutes. During the sham stimulation session, 2 mA of stimulation will be applied over the course of 90 sec, the electrodes will remain in place for the 30 minute duration.

SUMMARY:
Non-invasive brain stimulation has been shown to alter performance in both clinical and healthy populations on cognitive tasks. While the performance alterations have generally been shown to result in enhancement, mixed results remain in the literature. Much of the mixed results within the literature have been attributed to the use of different stimulation parameters, targeting of different brain areas, and using a variety of performance measures or assessing different constructs. However, non-invasive brain stimulation is a desirable method for enhancing Soldier performance given the ease of administration and minimal side effects as compared to other forms of performance enhancement (e.g., pharmaceuticals, caffeine). The objective of the current study is to evaluate the effects of non-invasive brain stimulation to the left dorsolateral prefrontal cortex in enhancing Soldier cognitive skills and performance on military tasks. A double blind within-subjects design will be used with healthy, rested Soldiers who will receive non-invasive brain stimulation and perform basic cognitive and operationally relevant tasks.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 (if active duty), 19 (if non-active duty) up to 40 years old.
2. Must have normal hearing, vision or corrected to normal vision, and cognitive function as determined by self-report and screening by study physician
3. Must have obtained at minimum 6 hours of sleep prior to data collection, as assessed by actigraphy data and self-report.
4. Must have refrained from consumption of caffeine, 16 hours, nicotine, 2 hours, and alcohol, 24 hours, prior to the study, assessed by self-report.

Exclusion Criteria:

1. The following medically-related exclusionary criteria will be used, as assessed and verified by the study physician:

   1. Haven taken any medications which induce drowsiness, such as over-the-counter antihistamines within 24 hours of participation in the study. Any self-medication will be assessed through self-report
   2. No current medical conditions or medications affecting cognitive function or attention.
   3. Any history of any attention deficit condition requiring medication.
   4. Any history of psychological/psychiatric disorder.
   5. Any history of seizures, migraines, or neurological disorders.
   6. History of a head injury involving loss of consciousness.
   7. Any metal implanted within the head (e.g., shrapnel, surgical clips) or any implanted devices (e.g., cardiac pacemaker, brain stimulator, hydrocephalic shunt).
   8. Skin condition on the scalp, such as psoriasis or eczema, or wounds on the head.
   9. Currently receiving hormonal therapy treatments, other than birth control or as determined by physicians.
   10. Potential for caffeine withdrawal symptoms that will impede cognitive testing.
2. Females with a known pregnancy, who test positively for pregnancy, or refuse the test will be excluded, given the lack of available research regarding the effects of tDCS during pregnancy. Known pregnancy will be assessed during screening, females without a known pregnancy will be requested to provide a urine sample during the screening procedures to ensure the absence of pregnancy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Military task performance | Folllowing stimulation; task lasts approximately 20 min
  Patrol exertion multitask
Military task performance | Folllowing stimulation; task lasts approximately 40 min
  Target acquisition
Cognitive function - Selective Attention | Approximately 3 minutes during stimulation
  Stroop test
Cognitive function - Multitasking/Working Memory | Approximately 5 minutes during stimulation
  Dual n-back
Cognitive function - Working Memory | Approximately 2 minutes during stimulation
  Digit span task
Cognitive function - Sustained attention | Approximately 7 minutes during stimulation
  Rapid Visual Information Processing Task
Cognitive function - Executive function | Approximately 2 minutes during stimulation
  Shifting Attention Task: Digit symbol substitution task

SECONDARY OUTCOMES:
Cognitive function - Impulsivity/Motor Control | Approximately 3 minutes after stimulation
  Stop signal task - response inhibition
Cognitive function - Risk Taking/ Decision Making | Approximately 1 minute after stimulation
  Delayed Discounting Task
Cognitive function - Cognitive Flexibility | Approximately 5 minutes after stimulation
  Uses Task

OTHER OUTCOMES:
Confounding factor - Sleepiness | Approximately 1 minute, before and after stimulation
  Karolinska Sleepiness Scale
Confounding factor - Circadian typology | Approximately 15 minutes during intake
  Morningness-Eveningness Questionnaire
Moderator variable - Intelligence | Approximately 15 minutes during intake
  Shipley's Institute of Living Scale
Moderator variable - Trait motivation | Approximately 10 minutes during intake
  Behavioral Avoidance/ Inhibition Scales
Side effects - mood symptoms | Approximately 3 minutes before and after stimulation
  Profile of Mood States - Short Form
Side effects - Physical side effects | Approximately 2 minutes before and after stimulation
  Symptom Checklist
Side effects - Physiology/health | Approximately 5 minutes before and after stimulation
  Welch Allyn Connex 6000

CONTACTS AND LOCATIONS:
Overall Officials: Katie Feltman, PhD, Principal Investigator — US Army Aeromedical Research Laboratory
Locations (1):
- U.S. Army Aeromedical Research Laboratory, Fort Rucker, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/33/NCT04155333/ICF_000.pdf